CLINICAL TRIAL: NCT02132793
Title: Remote Exercise for Learning Anger and Excitation Management (RELAX)
Brief Title: Remote Exercise for Learning Anger and Excitation Management
Acronym: RELAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pacific Islands Health Care System (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); Charles River Analytics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-12-C-0067
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2016-11

CONDITIONS: Anger; Stress Disorders, Post-Traumatic
Keywords: technology; mobile; anger management; anger; PTSD; veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Anger Management Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anger Management Therapy (Active Comparator): Anger Management Therapy (AMT) is a 12-session manual-driven cognitive-behavioral intervention found efficacious for anger management treatment.
  Interventions: Behavioral: Anger Management Therapy
- Anger Management Therapy & RELAX app (Experimental): Anger Management Therapy (AMT) is a 12-session manual-driven cognitive-behavioral intervention found efficacious for anger management treatment. RELAX app (1) enables the practice of anger management strategies remotely through mobile phone interfaces; (2) integrates with evidence-based treatments through implementing an existing CBT anger management course; (3) provides information, direction, and feedback through physiological sensors; and (4) supports communication and direction by the therapist through a web-based therapist interface and a remote and secure patient data server.
  Interventions: Behavioral: Anger Management Therapy & RELAX app

INTERVENTIONS:
Behavioral: Anger Management Therapy — Anger Management Therapy (AMT) is a 12-session manual-driven cognitive-behavioral intervention found efficacious for anger management treatment.
  Arms: Anger Management Therapy
Behavioral: Anger Management Therapy & RELAX app — Anger Management Therapy (AMT) is a 12-session manual-driven cognitive-behavioral intervention found efficacious for anger management treatment. RELAX app (1) enables the practice of anger management strategies remotely through mobile phone interfaces; (2) integrates with evidence-based treatments through implementing an existing CBT anger management course; (3) provides information, direction, and feedback through physiological sensors; and (4) supports communication and direction by the therapist through a web-based therapist interface and a remote and secure patient data server.
  Arms: Anger Management Therapy & RELAX app

SUMMARY:
The immediate objective of this project was to demonstrate the feasibility of Remote Exercises for Learning Anger and Excitation Management (RELAX). The application is a remote, technology- enabled, anger treatment and management system based on current evidence-based CBT interventions. The project's objective was to show that RELAX (1) enables the practice of anger management strategies remotely through mobile phone interfaces; (2) integrates with evidence-based treatments through the implementation of an existing CBT anger management course; (3) provides information, direction, and feedback through physiological sensors and signal analysis; and (4) supports communication and direction by the therapist through a web-based therapist interface.

DETAILED DESCRIPTION:
This project conducted a cognitive behavioral therapy (CBT) anger management treatment groups with a Veteran population using the RELAX application, collected weekly feedback from participants, and collaborate with the Sponsor to document initial efficacy, feasibility, and safety of the RELAX system. Outcome domains included: 1) clinical outcomes (symptom severity, social functioning); 2) process outcomes (perception of treatment, satisfaction, group therapy alliance, treatment compliance, and attrition and treatment credibility); and (3) Technical feasibility of the RELAX application. Study clinicians were 1) trained to conduct baseline and follow-up assessments 2) trained to conduct the standardized Anger Management Therapy (AMT) protocol at acceptable levels of adherence and competence and 3) trained how to use the technology and how to respond to technical difficulties. Study clinicians tested the feasibility of the RELAX application and showed that it can be integrated with CBT anger management therapies and support therapist communication through the technology.

ELIGIBILITY:
Inclusion Criteria:

* a score of 20 or higher on the 10-item Trait Scale of the STAXI
* participants taking psychoactive medications have to have a stable regimen for at least 45 days prior to study entry
* participants must be able to read, understand, and sign the consents themselves and be willing and able to comply with all study related procedures

Exclusion Criteria:

* active psychotic symptoms/disorder as determined by the Structured Clinical Interview (SCID) for Diagnostic and Statistical Manual of Mental Disorders(DSM)
* active homicidal or suicidal ideation as determined by the SCID
* any significant cognitive impairment or history of Organic Mental Disorder as determined by the SCID
* active (current) substance dependence as determined by the SCID (lifetime substance dependence or substance abuse not excluded)
* unwillingness to refrain from substance abuse during treatment
* female Veterans
* vulnerable persons such as those described in the section Ethical Considerations and Regulatory Issues, Vulnerable Population

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Dimensions of Anger Reactions (DAR-5) | up to 3 month follow-up
  The DAR-5 is a reliable and valid screening measure of common anger reactions. Its brevity is useful for rapidly assessing the presence of anger problems in different populations. The strength of the DAR-5 is that it employs a minimum number of items to measure the anger construct. Item content pertains to anger frequency, intensity, duration, interpersonal aggressiveness, and the extent to which anger interferes with interpersonal relationships.

SECONDARY OUTCOMES:
State-Trait Anger Expression Inventory-2 (STAXI-2) | Immediate post treatment and 3 month follow-up
  The STAXI-2 is a revised and expanded version of the original STAXI. The measure consists of items assessing the intensity of anger as an emotional state (State Anger) and the tendency of an individual to experience state anger, or anger proneness (Trait Anger). The Trait Anger scale measures individual differences in the disposition to experience anger. The Anger Expression scale provides an index of the frequency of anger expression. The STAXI has demonstrated strong reliability and validity.

OTHER OUTCOMES:
PTSD Checklist (PCL-5) | Immediate post treatment and 3 month follow-up
  The PCL will be used as an additional measure of PTSD symptoms. The PCL has been found to be a reliable and valid self-report measure of PTSD. Respondents indicate the degree to which they have been bothered by each of the 17 PTSD symptoms during the past month on a 5-point Likert scale, and item scores are summed.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret-Anne Mackintosh, Ph.D., Principal Investigator — VA Pacific Islands Healthcare System
Locations (1):
- VA Pacific Islands Healthcare System, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No